CLINICAL TRIAL: NCT04968509
Title: A Randomized Trial of PCSK9 Inhibitors in Calcific Aortic Valve Stenosis
Brief Title: Effect of PCSK9 Inhibitors on Calcific Aortic Valve Stenosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Principal Investigator, Zhi Jian Wang, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPISODE; 2022-2-1052 (Other Grant/Funding Number: Capital's Funds for Health Improvement and Research)
Record Dates: First submitted 2021-07-04; First posted 2021-07-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Aortic Stenosis
Keywords: PCSK9 Inhibitors; Calcific Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of | interventions — PCSK9 Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with PCSK9 inhibitors and conventional lipid-lowering therapy based on statins (Experimental): Patients in experimental group are treated with PCSK9 inhibitors (140mg with Evolocumab or 75mg with Alirocumab or 150mg with Tafolecimab subcutaneously every two weeks) and conventional lipid-lowering therapy based on statins (atorvastatin 20-40mg qd with or without ezetimibe 10mg qd, or rosuvastatin 10-20mg qd with or without ezetimibe 10mg qd).
  Interventions: Drug: PCSK9 inhibitors and statins with or without ezetimibe
- Treatment with only conventional lipid-lowering therapy based on statins (Other): Patients in control group are only treated with conventional lipid-lowering therapy based on statins (atorvastatin 20-40mg qd with or without ezetimibe 10mg qd, or rosuvastatin 10-20mg qd with or without ezetimibe 10mg qd).
  Interventions: Drug: Statins with or without ezetimibe

INTERVENTIONS:
Drug: PCSK9 inhibitors and statins with or without ezetimibe — Patients in experimental group are treated with PCSK9 inhibitors (140mg with Evolocumab or 75mg with Alirocumab or 150mg with Tafolecimab subcutaneously every two weeks) and conventional lipid-lowering therapy based on statins (atorvastatin 20-40mg qd with or without ezetimibe 10mg qd, or rosuvastatin 10-20mg qd with or without ezetimibe 10mg qd).
  Other Names: Proprotein convertase subtilisin/kexin type 9 inhibitors; Hydroxymethylglutaryl-Coenzyme A Reductase inhibitors; Ezetimibe
  Arms: Treatment with PCSK9 inhibitors and conventional lipid-lowering therapy based on statins
Drug: Statins with or without ezetimibe — Patients in control group are only treated with conventional lipid-lowering therapy based on statins (atorvastatin 20-40mg qd with or without ezetimibe 10mg qd, or rosuvastatin 10-20mg qd with or without ezetimibe 10mg qd).
  Other Names: Hydroxymethylglutaryl-Coenzyme A Reductase inhibitors; Ezetimibe
  Arms: Treatment with only conventional lipid-lowering therapy based on statins

SUMMARY:
Calcific aortic stenosis (CAS) can cause severe adverse cardiac events, but there are currently no effective drugs that can prevent or delay the progression of the disease. In fact, aortic valve replacement remains the only treatment option.

CAS has been shown to be associated with Lp(a), LDL-C and PCSK9. Several observational studies indicated that the use of statins to decrease LDL-C levels was associated with the reduced incidence of CAS, but no randomized controlled trials (RCTs) showd that statins had any benefit on the progression of CAS. This may be related to the limited reduction of LDL-C by statin therapy. The proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors have emerged as a new lipid-lowering drug. On the basis of statin therapy, PCSK9 inhibitors can further reduce LDL-C and Lp(a) levels by 50% to 60% and 20% to 30%, respectively. Some studies reported that elevated plasma PCSK9 levels were related to CAS and PCSK9 R46L loss-of-function mutation was associated with lower rates of CAS, and importantly, some observational studies found that PCSK9 inhibitors could reduce the incidence of CAS.

Our trial aims to investigate the effect of PCSK9 inhibitors on preventing or delaying the progression of CAS. A total of 160 patients with mild or moderate CAS or asymptomatic severe AS will be randomly assigned to receive either statins or PCSK9 inhibitors+statins. All patients will be followed for at least 2 years at 3, 6,9,12,15,18,21,24 months after randomization. Quality of life (EQ-5D-3L including the EUROQOL visual analogue scale) questionnaires were gathered during each visit. Echocardiography and computer tomography were performed and blood samples were withdrawn at baseline, at 2 years visit, and before withdrawal from the study.

The primary endpoint is the average annual change in peak aortic jet velocity on echocardiography. The secondary endpoints include average annual change in aortic valve area on echocardiography, average annual change in aortic valve calcification score on cardiac non-contrast computer tomography, heart valve surgery, change in quality-of-life scores, and average annual change in aortic and coronary artery calcification. Safety endpoints include all-cause death and cardiovascular events.

The results of this trial will provide a new idea for the treatment of patients with CAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with mild or moderate calcific aortic stenosis (peak aortic jet velocity ≥ 2m/s and < 4m/s or mean transvalvular gradients ≥ 20mmHg and < 40mmHg), or asymptomatic severe aortic stenosis (peak aortic jet velocity ≥ 4m/s or mean transvalvular gradients ≥ 40mmHg and no symptoms and/or signs related to aortic stenosis and negative exercise treadmill test)
* Patients who are required to be treated with a stable statin (atorvastatin or rosuvastatin) dose for at least 4 weeks and to have an LDL-C level of 80 mg/dL or higher or between 60 and 80 mg/dL (to convert LDL-C values to mmol/L, multiply by 0.0259) with 1 major or 3 minor cardiovascular risk factors. Major risk factors include atherosclerotic cardiovascular disease, myocardial infarction or hospitalization for unstable angina in the preceding 2 years, or type 2 diabetes mellitus. Minor risk factors include current cigarette smoking, hypertension, low levels of high-density lipoprotein cholesterol, family history of premature coronary heart disease, high sensitivity C-reactive protein (hsCRP) level of 2 mg/L or higher (to convert hsCRP values to nmol/L, multiply by 9.524), or age 50 years or older for men and 55 years or older for women
* Patients agree to participate in the study by signing an informed consent form

Exclusion Criteria:

* Any previous treatment with PCSK9 inhibitors
* Patients who must be treated with long-term PCSK9 inhibitors
* Patients who cannot maintain statin and/or PCSK9 inhibitor use for 24 months
* Hypersensitivity to PCSK9 inhibitors and/or statin
* Fasting triglyceride (TG) levels > 400mg/dL (4.5 mmol/L) at screening
* Thyroid hypofunction
* Active or chronic liver disease
* Severe renal dysfunction (eGFR < 30 ml/min/1.73m2)
* History of cerebral hemorrhage
* History of alcohol or drug abuse
* Known active infection, or major hematological, metabolic, or endocrine dysfunction
* Patients who have been treated with systemic steroids or cyclosporine within the past 3 months
* Active malignant tumor
* Any life-threatening condition with life expectancy less than 12 months
* Severe mitral stenosis (valve area<1cm2)
* Severe mitral or aortic regurgitation
* Patients who are scheduled to undergo heart valve surgery
* Left ventricular ejection fraction < 30% or severe heart failure (NYHA class III or IV)
* The presence of a permanent pacemaker or defibrillator
* Arrhythmias that are not controlled by drugs
* Child-bearing potential without contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The average annual change in peak aortic jet velocity | Up to 24 months
  The peak aortic jet velocity is measured by echocardiography.

SECONDARY OUTCOMES:
The average annual change in aortic valve area | Up to 24 months
  The aortic valve area is measured by echocardiography.
The average annual change in aortic valve calcification score | Up to 24 months
  The aortic valve calcification score is measured by cardiac noncontrast computer tomography.
Heart valve surgery | Up to 24 months
  Transcatheter aortic valve implantation or surgical aortic valve replacement
Change in quality-of-life scores | Up to 24 months
  Change in quality-of-life scores is assessed with the use of the EQ-5D-3L scale

OTHER OUTCOMES:
Safety endpoints | Up to 24 months
  All-cause death or cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Wang, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindman BR, Clavel MA, Mathieu P, Iung B, Lancellotti P, Otto CM, Pibarot P. Calcific aortic stenosis. Nat Rev Dis Primers. 2016 Mar 3;2:16006. doi: 10.1038/nrdp.2016.6. PMID 27188578
- [Background] Rajamannan NM, Evans FJ, Aikawa E, Grande-Allen KJ, Demer LL, Heistad DD, Simmons CA, Masters KS, Mathieu P, O'Brien KD, Schoen FJ, Towler DA, Yoganathan AP, Otto CM. Calcific aortic valve disease: not simply a degenerative process: A review and agenda for research from the National Heart and Lung and Blood Institute Aortic Stenosis Working Group. Executive summary: Calcific aortic valve disease-2011 update. Circulation. 2011 Oct 18;124(16):1783-91. doi: 10.1161/CIRCULATIONAHA.110.006767. No abstract available. PMID 22007101
- [Background] Smith JG, Luk K, Schulz CA, Engert JC, Do R, Hindy G, Rukh G, Dufresne L, Almgren P, Owens DS, Harris TB, Peloso GM, Kerr KF, Wong Q, Smith AV, Budoff MJ, Rotter JI, Cupples LA, Rich S, Kathiresan S, Orho-Melander M, Gudnason V, O'Donnell CJ, Post WS, Thanassoulis G; Cohorts for Heart and Aging Research in Genetic Epidemiology (CHARGE) Extracoronary Calcium Working Group. Association of low-density lipoprotein cholesterol-related genetic variants with aortic valve calcium and incident aortic stenosis. JAMA. 2014 Nov 5;312(17):1764-71. doi: 10.1001/jama.2014.13959. PMID 25344734
- [Background] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002
- [Background] Rajamannan NM, Subramaniam M, Springett M, Sebo TC, Niekrasz M, McConnell JP, Singh RJ, Stone NJ, Bonow RO, Spelsberg TC. Atorvastatin inhibits hypercholesterolemia-induced cellular proliferation and bone matrix production in the rabbit aortic valve. Circulation. 2002 Jun 4;105(22):2660-5. doi: 10.1161/01.cir.0000017435.87463.72. PMID 12045173
- [Background] Weiss RM, Ohashi M, Miller JD, Young SG, Heistad DD. Calcific aortic valve stenosis in old hypercholesterolemic mice. Circulation. 2006 Nov 7;114(19):2065-9. doi: 10.1161/CIRCULATIONAHA.106.634139. Epub 2006 Oct 30. PMID 17075015
- [Background] Cowell SJ, Newby DE, Prescott RJ, Bloomfield P, Reid J, Northridge DB, Boon NA; Scottish Aortic Stenosis and Lipid Lowering Trial, Impact on Regression (SALTIRE) Investigators. A randomized trial of intensive lipid-lowering therapy in calcific aortic stenosis. N Engl J Med. 2005 Jun 9;352(23):2389-97. doi: 10.1056/NEJMoa043876. PMID 15944423
- [Background] Chan KL, Teo K, Dumesnil JG, Ni A, Tam J; ASTRONOMER Investigators. Effect of Lipid lowering with rosuvastatin on progression of aortic stenosis: results of the aortic stenosis progression observation: measuring effects of rosuvastatin (ASTRONOMER) trial. Circulation. 2010 Jan 19;121(2):306-14. doi: 10.1161/CIRCULATIONAHA.109.900027. Epub 2010 Jan 4. PMID 20048204
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Bergmark BA, O'Donoghue ML, Murphy SA, Kuder JF, Ezhov MV, Ceska R, Gouni-Berthold I, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Gaciong Z, Lewis BS, Schiele F, Jukema JW, Pedersen TR, Giugliano RP, Sabatine MS. An Exploratory Analysis of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibition and Aortic Stenosis in the FOURIER Trial. JAMA Cardiol. 2020 Jun 1;5(6):709-713. doi: 10.1001/jamacardio.2020.0728. PMID 32347887
- [Background] Capoulade R, Cariou B. Editorial commentary: Lp(a) and calcific aortic valve stenosis: Direct LPA targeting or PCSK9-Lowering therapy? Trends Cardiovasc Med. 2021 Jul;31(5):312-314. doi: 10.1016/j.tcm.2020.06.009. Epub 2020 Jul 2. No abstract available. PMID 32623063
- [Background] Poggio P, Songia P, Cavallotti L, Barbieri SS, Zanotti I, Arsenault BJ, Valerio V, Ferri N, Capoulade R, Camera M. PCSK9 Involvement in Aortic Valve Calcification. J Am Coll Cardiol. 2018 Dec 18;72(24):3225-3227. doi: 10.1016/j.jacc.2018.09.063. No abstract available. PMID 30545459
- [Background] Perrot N, Valerio V, Moschetta D, Boekholdt SM, Dina C, Chen HY, Abner E, Martinsson A, Manikpurage HD, Rigade S, Capoulade R, Mass E, Clavel MA, Le Tourneau T, Messika-Zeitoun D, Wareham NJ, Engert JC, Polvani G, Pibarot P, Esko T, Smith JG, Mathieu P, Thanassoulis G, Schott JJ, Bosse Y, Camera M, Theriault S, Poggio P, Arsenault BJ. Genetic and In Vitro Inhibition of PCSK9 and Calcific Aortic Valve Stenosis. JACC Basic Transl Sci. 2020 Jul 1;5(7):649-661. doi: 10.1016/j.jacbts.2020.05.004. eCollection 2020 Jul. PMID 32760854
- [Derived] Zheng Y, Li Q, Yang Y, Yang J, Liu Z, Ma X, Wang Z. Rationale and Design of the EPISODE Trial: A Randomized Controlled Trial on the Effect of PCSK9 Inhibitors in Calcific Aortic Valve Stenosis. J Am Heart Assoc. 2025 Oct 7;14(19):e042112. doi: 10.1161/JAHA.125.042112. Epub 2025 Sep 19. PMID 40970544